CLINICAL TRIAL: NCT02438657
Title: Ultrasound-guided Median Nerve Block With Dextrose 5% Hydrodissection: Determination of the Minimal Effective Volume of Local Anesthetic
Brief Title: Ultrasound-guided Nerve Block: Determination of the Minimal Effective Volume of Local Anesthetic
Acronym: VMAL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014/07; 2014-000571-50 (EudraCT Number)
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Surgery
MeSH Terms: interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: Ascending dose model
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- median nerve block (Experimental): An ultrasound-guided nerve block with dextrose 5% hydrodissection is performed in each case. The first patient will receive a 2 mL local anesthetic solution. For following patients, the volume of local anesthetic depends on the clinical result of the previous patient:
  * increase of the volume (0.5 mL) in case of failure,
  * no change or decrease (0.5 mol) in case of success; a randomization is made in this case (BCD method, Stylianou M, Flournoy N. Dose finding using the biased coin up-and-down design and isotonic regression. Biometrics 2002;58:171-7)
  Interventions: Procedure: median nerve block

INTERVENTIONS:
Procedure: median nerve block
  Other Names: lidocaine with epinephrine (20 mg/ml)

SUMMARY:
Ultrasound guidance can reduce the required local anesthetic volume for successful peripheral nerve block.

The aim of the study is to determine the minimum volume of local anesthetic to achieve an ultrasound-guided median nerve block with a dextrose 5% hydrodissection approach.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years from 18 to 80 years with an ASA (American Society of Anesthesiologists) physical status I-II
* elective hand ambulatory surgery with a maximum duration of 30 minutes involving the median nerve and performed with elbow nerve blocks

Exclusion Criteria:

* pregnant or lactating women,
* contra-indication to regional anesthesia
* diabetes mellitus,
* effective anticoagulation or antiplatelet therapy, laboratory evidence of abnormal bleeding
* neurological disease ( including carpal tunnel syndrome or neuromuscular disease detected by preoperative neurological examination in the median nerve)
* infection at the puncture site
* contra-indication to the administration of lidocaine, notably allergy
* contra-indication to the administration of lidocaine with epinephrine
* not speaking French

Exclusion from the study:

* patient having an intraneural injection of the median nerve defined by swelling appearance are excluded from analysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Minimal effective volume of local anesthetic | 1 hour
  Effective volume of local anesthetic to obtain a successful median nerve block block in 95% of patients defined as complete light touch block at the palmar aspect of the 2 distal phalanges of the index finger during a 30 minute evaluation period (mL)

SECONDARY OUTCOMES:
Nerve block onset time | 1 hour
  Onset time for complete cold light touch and motor block at 30 min and 45 min.
Success rate of the median nerve block | 1 hour
  Success rate concerns:
  * success rate of sensitive block: complete cold and light touch block at 30 min and 45 min at the palmar aspect of the 2 distal phalanges of the index finger and on the thenar eminence
  * success rate of motor block: complete motor block at 30 min and 45 min
Additional local anesthetic | 2 hours
  * Percentage of cases where additional local anesthetic was necessary before the incision (%), i.e; performed by anesthesiologist
  * Percentage of cases where additional local anesthetic was necessary after the incision (%), i.e; performed by surgeon
Duration of analgesia | 1 day
  Time to first analgesic requirement (minutes)
Duration of the block | 1 day
  Delay between the completion of the block and the returned to normal onset of sensory and motor recovery of the first three fingers of the hand) (minutes)
Complications | 1 month
  * complications occurring during the procedure (pain, paresthesia, intraneural injection and vascular puncture),
  * complications noticed at the first postoperative month (residual pain, paresthesia, dysesthesia, weakness)
Block procedure time | One hour
  Time taken to perform hydrodissection with dextrose 5% and inject the local anesthetic (min)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Dufour, MD, Principal Investigator — Centre Hospitalier de la Côte Basque, 64100 Bayonne, France
Locations (2):
- France (2):
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Hopital privé de l'Ouest Parisien, Trappes

REFERENCES:
- [Derived] Dufour E, Jaziri S, Novillo MA, Aubert L, Chambon A, Kutz R, Vallee A, Fischler M. A randomized trial to determine the minimum effective lidocaine volume for median nerve block using hydrodissection. Sci Rep. 2022 Jan 7;12(1):52. doi: 10.1038/s41598-021-03660-7. PMID 34996918